CLINICAL TRIAL: NCT03839537
Title: Exposure of Taxi Drivers to Ultrafine Particles and Black Carbon Within Their Vehicles: Determinants of In-vehicle Exposure and Short Term Respiratory Impact.
Brief Title: Exposure of Taxi Drivers to Ultrafine Particles and Black Carbon Within Their Vehicles
Acronym: PUF-TAXI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); Centre national de la recherche scientifique - Lebanon (CNRS-L) (Unknown); French Environment and Energy Management Agency (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: K180303J; 2018-A00811-54 (Other: ID-RCB)
Record Dates: First submitted 2019-01-07; First posted 2019-02-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Ventilation
Keywords: Ultrafine particles; black carbon; taxi drivers; respiratory function test; occupational exposure
MeSH Terms: interventions — Skin Tests; Patch Tests; Spirometry; Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure measurement — * 2 measurements per subject (in warm season and in cold season)
  * Devices placed inside taxi vehicles on the passenger seat in a sampling bag
  Other Names: Exposure measurement of UFP, BC, NO2, CO, CO2
Other: Spirometry test — * 2 measurements per subject - before and after the work shift - in warm and cold seasons
  * Subject will inhale and exhale in the device
  Other Names: Spirobank II
Diagnostic Test: Exhaled carbon monoxide test — * 2 measurements per subject - before and after the work shift - in warm and cold seasons
  * Subject will exhale in the device
  Other Names: Smokerlyzer- Micro
Diagnostic Test: Skin allergy test — - Performed by a physician during the inclusion clinical examination
  Other Names: Prick test
Diagnostic Test: Spirometry test — - Performed by a physician during the inclusion clinical examination
Diagnostic Test: Fractional Exhaled Nitric Oxide Testing — - Performed by a physician during the inclusion clinical examination

SUMMARY:
Brief Summary Short description of the protocol intended for the lay public. Include a brief statement of the study hypothesis. (Limit: 5000 characters)

Example: The purpose of this study is to determine whether prednisone, methotrexate, and cyclophosphamide are effective in the treatment of rapidly progressive hearing loss in both ears due to autoimmune inner ear disease (AIED). This project is part of a research field on the role, not yet fully understood, of atmospheric pollution, especially from road traffic, on respiratory health and allergies, particularly on the development / onset of symptoms and functional disturbances. The ultrafine fraction of particles (UFPs - particles smaller than 100 nm in diameter) is of recent interest because of their ability to induce inflammatory effects, oxidative stress and may contribute to the exacerbation of asthma symptoms in susceptible individuals. UFPs, with their high number concentration and surface area and their small diameter are able not only to convey other contaminants, but also to contribute to a high deposition efficiency, into the alveoli in the lungs. Recently it appeared relevant to be interested in black carbon (BC), components of PM2.5 (particulate matter with a diameter less than 2.5 micrometers), suspected of being responsible for their toxicity. Current epidemiological knowledge of the effects of UFPs and BC are few as compared to those on fine particles. Some professionals, such as police, drivers (taxis, truckers ...), delivery men, postal workers, workers on roads and highways, etc. are heavily exposed, during their working hours, to air pollution due to road traffic. These occupational groups appear to be at greater risk for developing respiratory, cardiovascular and neurological diseases than the general population. Occupational exposure to diesel exhaust has been associated with an increased risk of lung cancer mortality and chronic obstructive pulmonary disease. Occupational exposure to UFPs and BC has rarely been measured due to a lack of suitable devices. Therefore, this project's originality consists in measuring UFPs and BC by using portable devices developed in the recent years. The use of these devices, linking their recordings with ventilatory measures and repeating them, offers the rare opportunity to study the short-term respiratory health impact of this occupational exposure, which has never been described in the literature. Our research aims to: 1/ quantify the occupational exposure of taxi drivers to UFP, BC, oxides of carbon (CO, CO2) and to nitrogen dioxide (NO2), 2/ identify spatio-temporal variability and patterns of exposure related to occupational tasks, 3/ study the impact of this occupational exposure to UFP and BC on ventilation performances and respiratory symptoms.

DETAILED DESCRIPTION:
The study is based on a random sampling of 100 taxi drivers, working full-time day shift, in Paris, members of three Trade Unions. It will be conducted over a period of two years in warm and cold season. The research will begin with an inclusion clinical examination. It consists on determining the overall health status of the participants by administering a standardized questionnaire and performing spirometry test, prick test and FENO measurement. The exposure assessment will be based on continuous measurement of UFP, BC, carbon monoxide (CO) and NO2, by portable devices during a working day (± 11 hours). On the same day, two spirometry tests and two measurements of exhaled carbon monoxide will be performed at the beginning and at the end of the shift, using handheld devices. Multivariate analysis will provide spatio-temporal distributions of individual exposures and their determinants. Generalized Estimating Equations (GEE) multivariate models will be used to determine the relation between exposure (UFP, BC) and respiratory symptoms, ventilation performances, adjusting for potential confounding/modifying factors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Full time licensed taxi driver
* Subjects with more than 6 months of job tenure (as a taxi driver)
* Subjects affiliated to a social security scheme
* Subjects must have signed an informed consent and are willing to participate in the study

Exclusion Criteria:

* Subjects having difficulty to understand the French language
* Subjects with less than 6 months of job tenure (as a taxi driver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Mean number of ultrafine fraction of particles (UFP) | 6 months
  per cm3 of air [from 1000 to 1000000 particles (pt)/cm3] - 8-11 h recording on 1 working day for each subject - repeated measurement in cold and warm seasons (6 months apart)
Mean concentration of black carbon (BC) | 6 months
  measurement of BC exposure concentrations per cubic meter (ng/m3) by the microAeth AE51 - 8-11 h recording on 1 working day for each subject - repeated measurement in cold and warm seasons (6 months apart)
Difference between the values of the forced vital capacity (FVC) measured before and after work shift | 36 months
  measurement of FVC in liters by a portable spirometer before and after the work shift according to procedures described by The European Respiratory Society and the American Thoracic Society (2005) - 2 measurements per subject - before and after the work shift - 1 working day Repeated measurement in cold and warm seasons (6 months apart) Overall period: 2 working days (one in each season) - 36 months
Difference between the values of the forced expiratory volume in one second (FEV1) measured before and after work shift | 36 months
  measurement of FEV1 in liters by a portable spirometer before and after the work shift according to procedures described by The European Respiratory Society and the American Thoracic Society (2005) -2 measurements per subject - before and after the work shift - 1 working day Repeated measurement in cold and warm seasons (6 months apart) Overall period: 2 working days (one in each season) - 36 months
Difference between the values of the forced expiratory flow between 25 and 75 % of FVC (FEF25-75) measured before and after work shift | 36 months
  measurement of FEF25-75 in liters by a portable spirometer before and after the work shift according to procedures described by The European Respiratory Society and the American Thoracic Society (2005). -2 measurements per subject - before and after the work shift - 1 working day Repeated measurement in cold and warm seasons (6 months apart) Overall period: 2 working days (one in each season) - 36 months
Difference between the rates of the peak expiratory flow (PEF) measured before and after work shift | 36 months
  measurement of PEF in liter per second (L.s-1) by a portable spirometer before and after the work shift according to procedures described by The European Respiratory Society and the American Thoracic Society (2005)-2 measurements per subject - before and after the work shift - 1 working day Repeated measurement in cold and warm seasons (6 months apart) Overall period: 2 working days (one in each season) - 36 months
Acute respiratory symptoms through self-administered questionnaire | 36 months
  by means of a self-completion questionnaire, participants report their acute respiratory symptoms felt during the measurement day - Reported before and after the work shift per subject - In cold and warm seasons (6 months apart)- Overall period: reported during 2 working days (one in each season) - 36 months

SECONDARY OUTCOMES:
Characteristics of vehicles recorded by a self-administered questionnaire | 36 months
  fuel, age and type of the vehicle, air conditioning, air cabin filter reported by a self-administered questionnaire - after the work shift per subject - In cold and warm seasons (6 months apart) Overall period: reported during 2 working days (one in each season) - 36 months
Characteristics of the trips recorded by a self-administered questionnaire | 36 months
  speed, opened/closed windows, smoking, breaks, etc. reported by a self-administered questionnaire - after the work shift per subject - In cold and warm seasons (6 months apart) Overall period: reported during 2 working days (one in each season) - 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynda BENSEFA-COLAS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Paris Descartes University, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hachem M, Saleh N, Bensefa-Colas L, Momas I. Determinants of ultrafine particles, black carbon, nitrogen dioxide, and carbon monoxide concentrations inside vehicles in the Paris area: PUF-TAXI study. Indoor Air. 2021 May;31(3):848-859. doi: 10.1111/ina.12779. Epub 2020 Dec 22. PMID 33350528